CLINICAL TRIAL: NCT04632004
Title: Questionnaire Regarding the Effect of Wearing Face Masks on Oral Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, PD Dr. med. dent., Dr. rer. medic., Senior Dental Practitioner, University Medical Center Goettingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FaceMasks-OralHealth; 28/10/20 (Other: Local Ethics Commission)
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Dry Mouth; Halitosis
MeSH Terms: conditions — Xerostomia; Halitosis

STUDY DESIGN:
Intervention Model Description: Patients, visitors, and staff members of the University Medical Center Goettingen are invited to participate within the survey study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaire survey (Other): Patients, visitors, and staff members of the University Medical Center Goettingen are invited to participate within our survey study. Study participation has no effect on any medical treatment.
  Interventions: Other: Invitation to participate

INTERVENTIONS:
Other: Invitation to participate — Patients, visitors, and staff members of the University Medical Center Goettingen are invited to participate within our survey study. Study participation has no effect on any medical treatment.

SUMMARY:
During the current COVID-19 pandemic, the use of face masks is recommended / mandatory to prevent infection. Patients and students have reported to experience limitations in their oral health-related quality of life, especially with regard to the occurrence of dry mouth and halitosis, while wearing face masks.

Scientific studies regarding the effects of face masks have so far focused exclusively on medical staff. Studies among the general population are not yet available, but are of interest as dry mouth is a risk factor for dental diseases (e.g., caries, erosion).

Therefore, the present study aims at performing a questionnaire survey regarding self-perceived dry mouth and halitosis and the use of face masks (type, wearing time).

ELIGIBILITY:
Inclusion Criteria:

* Patients, visitors, and staff members of the University Medical Center Goettingen

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3750 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Self-perceived dry mouth | During the 1 day of questionnaire survey
  Questionnaire items based on the shortened Xerostomia Inventory
Self-perceived halitosis | During the 1 day of questionnaire survey
  Questionnaire items

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Goettingen, Dept. of Preventive Dentistry, Periodontology and Cariology, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farronato M, Boccalari E, Del Rosso E, Lanteri V, Mulder R, Maspero C. A Scoping Review of Respirator Literature and a Survey among Dental Professionals. Int J Environ Res Public Health. 2020 Aug 17;17(16):5968. doi: 10.3390/ijerph17165968. PMID 32824564
- [Background] Rebmann T, Carrico R, Wang J. Physiologic and other effects and compliance with long-term respirator use among medical intensive care unit nurses. Am J Infect Control. 2013 Dec;41(12):1218-23. doi: 10.1016/j.ajic.2013.02.017. Epub 2013 Jun 12. PMID 23768438
- [Background] Shenal BV, Radonovich LJ Jr, Cheng J, Hodgson M, Bender BS. Discomfort and exertion associated with prolonged wear of respiratory protection in a health care setting. J Occup Environ Hyg. 2012;9(1):59-64. doi: 10.1080/15459624.2012.635133. PMID 22168256
- [Result] Kanzow P, Dylla V, Mahler AM, Hrasky V, Rodig T, Barre F, Scheithauer S, Wiegand A. COVID-19 Pandemic: Effect of Different Face Masks on Self-Perceived Dry Mouth and Halitosis. Int J Environ Res Public Health. 2021 Aug 31;18(17):9180. doi: 10.3390/ijerph18179180. PMID 34501768